CLINICAL TRIAL: NCT05315453
Title: Brief Telehealth Cognitive Rehabilitation Following Mild Traumatic Brain Injury: A Pilot Study
Brief Title: Brief Telehealth Cognitive Rehabilitation Following Mild TBI
Acronym: On-TRACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Pagulayan, Associate Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00013494
Record Dates: First submitted 2021-12-13; First posted 2022-04-07 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Mild Traumatic Brain Injury; Cognitive Impairment
MeSH Terms: conditions — Brain Concussion; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Cognitive Rehabilitation (Experimental): 5-session Cognitive Rehabilitation intervention administered over telehealth
  Interventions: Behavioral: Brief Cognitive Rehabilitation

INTERVENTIONS:
Behavioral: Brief Cognitive Rehabilitation — 5-session Cognitive Rehabilitation intervention that can be administered over telehealth.

SUMMARY:
In the United States, more than a million people sustain a mild traumatic brain injury (mTBI) every year. Although many recover fully, emerging literature suggests a high number of individuals report chronic, and functionally disabling, cognitive difficulties. Among Veterans, a nationwide survey found that more than 75% of 55,000 Veterans with a history of mTBI reported persistent moderate to severe levels of forgetfulness and poor concentration.

Reduced cognitive functioning following mTBI contributes to significant functional impairment, including underemployment, relationship difficulties, and reduced community integration for years post injury. Despite the significant individual and societal impact, evidence to guide interventions and treatment for this population remains limited. Even more limited are validated telehealth options for these symptoms, a critical means by which access to care can be improved, especially during the COVID-19 pandemic. The proposed pilot study will address this gap by evaluating the feasibility, acceptability, and preliminary effectiveness of a brief (5-session) cognitive rehabilitation intervention that was developed for individuals with mTBI and that will be administered over video-based telehealth technology. The development of this intervention was supported by a grant from the Department of Defense, with critical elements identified through surveys completed by clinicians and veterans with a history of mTBI, and also the clinical expertise of the team.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+;
* Read, speak, understand English;
* History of at least one mTBI;
* Endorses moderate to severe cognitive difficulties in one or more of Neurobehavioral Symptom Inventory items M-P;
* Ability and willingness to participate in audio recorded sessions over video telehealth platform in a private setting, including equipment and internet access;
* Lives within 2 hours of VA Puget Sound or affiliated clinics/University of Washington;
* Will be in Washington State when engaging in treatment sessions

Exclusion Criteria:

* Significant cognitive impairment that would limit ability to engage on treatment;
* Neurologic injury or illness that affects cognitive functioning, including history of moderate or severe TBI;
* History of TBI in the past 3 months, from the date of screening;
* History of serious mental illness involving psychotic symptoms;
* Current psychotic or manic symptoms;
* Current or active flag, or documentation in medical record, for behavior or suicide risk;
* Current (within the past 3 months) Substance Use Disorder (not including caffeine or nicotine disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of administering the On-TRACC intervention to individuals with mTBI | At the completion of 5 week intervention
  Feasibility measures will include rate of enrollment of eligible individuals as well as dropout rate for enrolled participants. We will also evaluate participant adherence, including proportion of treatment sessions attended and number of days that homework was completed.

SECONDARY OUTCOMES:
Participant satisfaction with On-TRACC intervention | End of each treatment session and at treatment completion, 5 weeks total.
  Participants will provide feedback on individual treatment sessions and at the end of treatment regarding intervention content. Participants will complete a Weekly Therapy Rating form after each treatment session and an End of Treatment Patient Feedback Form at the end of treatment to provide satisfaction ratings.
Preliminary effectiveness of On-TRACC intervention in decreasing post-concussive symptoms | Baseline (pre-treatment) and at the end of the 5-week On-TRACC intervention, 5 week time-frame on average
  Pre-post treatment change in post-concussive symptoms (Neurobehavioral Symptom Inventory) will be evaluated.
Preliminary effectiveness of On-TRACC intervention at decreasing self-reported cognitive difficulties | Baseline (pre-treatment) and at the end of the 5-week On-TRACC intervention, 5 week time-frame on average
  Pre-post treatment change in self-reported cognitive difficulties (NeuroQol Item Bank Cognitive Function SF) will be evaluated.
Preliminary effectiveness of On-TRACC intervention at improving self-efficacy | Baseline (pre-treatment) and at the end of the 5-week On-TRACC intervention, 5 week time-frame on average
  Pre-post treatment change in self-efficacy (Cognitive Concerns Self-Efficacy Scale) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pagulayan, PhD, Principal Investigator — VA Puget Sound Health Care System/University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No